CLINICAL TRIAL: NCT03464201
Title: Open Label Phase II Clinical Trial of Enzalutamide in Metastatic or Advanced Non-resectable Granulosa Cell Ovarian Tumors: GreKo III Study
Brief Title: Enzalutamide in Metastatic or Advanced Non-resectable Granulosa Cell Ovarian Tumors: GREKO III Study
Acronym: GREKO III
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Tumores Huérfanos e Infrecuentes (Other)
Collaborators: Astellas Pharma Inc (Industry); Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GETHI 2016-01; 2015-004469-10 (EudraCT Number)
Record Dates: First submitted 2018-02-19; First posted 2018-03-13 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enzalutamide (Experimental): Enzalutamide 160 mg daily p.o. (4 capsules 40mg per day)
  Interventions: Drug: Enzalutamide 40 MG

INTERVENTIONS:
Drug: Enzalutamide 40 MG — Enzalutamide 160 mg p.o. every day

SUMMARY:
The good tolerability profile of enzalutamide, the fact that the administration of steroids is not necessary and the impressive results achieved in prostate cancer, make this drug an ideal candidate to be tested in ovarian granulosa cancer, a tumor that could somehow be considered as "female prostate cancer".

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given written informed consent
* Women aged 18 years or over
* Eastern Cooperative Oncology Group (ECOG) ≤ 1
* Diagnosis of histologically confirmed ovarian granulose carcinoma
* Availability of sufficient biopsy material for confirmation of the diagnosis by a centralized pathologist and determination of the mutation FOXL2402C→ G(C134W). If this material is not available, principal investigator of the study will confirm eligibility of the patient.
* Metastatic or unresectable disease
* Radiologically measurable disease. In case you there is not measurable disease, principal investigator of the study will confirm eligibility of the patient. - - Life expectancy ≥ 12 weeks
* Patients with adequate hepatic function, defined by: Aspartate transaminase (AST) and alanine aminotransferase (ALT) serum values ≤ 3 x upper limit of normal (except in the presence of metastasis in which case values ≤ 5 x upper limit of normal will be allowed), Total bilirubin values ≤ 1,5 x upper limit of normal
* Patients with adequate bone marrow function, defined by: Absolute neutrophil count ≥ 1.5 x 109 / L, Platelets ≥100 x 109/L, Hemoglobin ≥ 9 g/dL
* Patients with adequate renal function: serum creatinine ≤ 1,5 x upper limit of normal
* Absence of any disability to follow the study protocol
* Women childbearing potential who are sexually active, not undergoing hysterectomy or double adnexectomy, should follow the following contraceptive indications: Negative Pregnancy Test in serum or urine in the 72 hours before the start of treatment, use of a medically accepted method of contraception during: 2 months prior to the start of study treatment, during the study and up to 3 months after the last dose of treatment.

Exclusion Criteria:

* Patients with another primary tumor 2 years before beginning the drug under study, with the exception of adequately treated or totally surgically removed cervical carcinoma in-situ or basalioma or superficial bladder carcinoma
* Patients who have received radical radiotherapy ≤ 4 weeks prior to the start of study treatment or who have not recovered from toxicities of radiotherapy. Palliative radiation therapy for painful bone lesions bone is allowed up to 14 days prior to the beginning of the study treatment
* History of seizures or any conditions that may predispose to suffer them
* Current or previously treated brain metastases or disease leptomeningeal.
* Patients with cardiac insufficiency or heart disease clinically significant including any of the following: History or presence of uncontrolled severe ventricular arrhythmias, clinically significant resting bradycardia, any of the following diseases within 6 months prior to the start of the study drug -Myocardial infarction (MI), severe or unstable angina, coronary revascularization, congestive cardiac insufficiency (CCI), cerebrovascular accident (CVA), transient ischemic accident (TIA)-
* Patients with altered gastrointestinal function or with gastric disease that significantly alters the absorption of enzalutamide, such as for example: severe ulcer diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, extensive resection (> 1m) of the small bowel or inability to swallow oral medication. The previous partial or total gastrectomy is not an exclusion criterion.
* Diagnosis of human immunodeficiency virus (HIV) infection.
* Pregnant or lactating women.
* Women of childbearing potential not using an effective contraceptive method. - Patients who do not want or can follow the study protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Due to kind of disease only female patients are acceptable for the trial
Enrollment: 16 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 6 months
  Number of responses according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Clinical benefit rate | Up to 6 months
  Stabilization of disease plus the sum of partial and complete responses according to RECIST 1.1 criteria.
Progression-free survival (PFS) | Up to 6 months
  Number of progression of the disease according to RECIST 1.1 criteria or death of the patient for any cause
Overall survival (OS) | Up to 6 months
  Number of deaths for any cause.
Incidence of Treatment-Emergent Adverse Events | Up to 6 months
  Number of Adverse Events per patient

CONTACTS AND LOCATIONS:
Overall Officials: Garcia-Donas, MD, Principal Investigator — CIOCC (Hospital Universitario HM Sanchinarro)
Locations (8):
- Spain (8):
  - Hospital de Mar, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Hospital Madrid Sanchinarro (CIOCC), Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital de Navarra, Pamplona
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia-Donas J, Redondo A, Santaballa A, Garrigos L, Rubio MJ, Lainez N, Gonzalez MI, Cueva JF, Barquin A, Grazioso TP, Hurtado A, Sevillano E, Grande E, Rodriguez-Moreno JF, Navarro P. Phase II clinical trial assessing the efficacy of enzalutamide in advanced non-resectable granulosa cell ovarian tumors: The GREKO III study (GETHI2016-01). Gynecol Oncol. 2024 Dec;191:233-239. doi: 10.1016/j.ygyno.2024.10.019. Epub 2024 Oct 24. PMID 39454227